CLINICAL TRIAL: NCT00741910
Title: Extension Study of CNI-1493 for Treatment of Moderate to Severe Crohn's Disease
Brief Title: Extension Study of Semapimod 60 mg IV x 3 Days
Acronym: CD06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNI-1493-CD06
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2012-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; TNF-alpha inhibitor; MAP Kinase inhibitor; CNI-1493
MeSH Terms: conditions — Crohn Disease | interventions — semapimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Semapimod 60 mg IV q 6 - 10 weeks
  Interventions: Drug: Semapimod

INTERVENTIONS:
Drug: Semapimod — semapimod IV 60 mg x 3 days q 6 - 10 weeks
  Other Names: CNI-1493

SUMMARY:
Study CNI-1493-CD06 is an open, single-arm extension studies to CD03 and CD05. CDAI is the only efficacy measure assessed in this study. The safety of multiple courses of semapimod is to be determined by the incidence of clinical and laboratory adverse events.

ELIGIBILITY:
Inclusion Criteria:

The study was open to patients who had satisfactorily completed either study CNI-1493-CD-03 or CNI-1493-CD-05. Initial entry criteria were:

1. Patients who satisfactorily completed either study CNI-1493-CD-03 or CD-05 were eligible for participation in this study. Satisfactory completion was defined as follows:

   1. The patient completed 5 treatment courses in the previous trial.
   2. The patient had responded to treatment, as defined by a decrease in CDAI of at least 70 points from original baseline (prior to treatment on study CD-02 or CD-04) at the last assessment for study CD-03 or CD-05, respectively. The decrease had to be attributable to semapimod treatment. Thus, patients whose response was attributable to other anti-Crohn's disease therapy are not to be included.
   3. The patient had no adverse event >grade 2 felt to be probably or definitely related to study medication.
   4. The patient did not meet any discontinuation criterion in previous trial.
2. Patients had to sign informed consent specifically for this study, in addition to the consents for the previous studies, CNI-1493-CD-02 or CD-03, and CNI-1493-CD-04 or CD-05.
3. Patients could not take any other investigational therapies during the course of this study.
4. Men and women of childbearing potential had to be using a barrier method (diaphragm or condom) of contraception and continue doing so for at least 3 months after last study medication. It was strongly recommended that two forms be used.
5. Patients had to be able to adhere to the study visit schedule and/or protocol requirements.

Exclusion Criteria:

Could not have met any of the exclusion criteria for the CD02, 03, 04 or 05 studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index (CDAI) | Every 6 - 10 weeks

SECONDARY OUTCOMES:
Safety | Every 6 - 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daan Hommes, MD, Principal Investigator — Academic Medical Center, Netherlands
Locations (8):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Long Island Clinical Research Associates, Great Neck, New York
  - Asher Kornbluth, MD, New York, New York
- Benjamin Franklin University, Berlin, Germany
- Israel (3):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Hospital, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Erasmus Medical Center, Rotterdam, Netherlands